CLINICAL TRIAL: NCT00343811
Title: A 6-week, Double-Blind, Placebo-Controlled, Parallel Group Randomized Withdrawal Study to Evaluate the Continued Efficacy of Modafinil Treatment in Dosages up to 425mg/Day in Patients With Attention-Deficit/Hyperactivity Disorder Who Are Responders to Modafinil Treatment, Followed by a 12-Month Open-Label Extension Period
Brief Title: Study to Evaluate the Efficacy of Modafinil Treatment in Patients With Attention Deficit Hyperactivity Disorder (ADHD) Who Are Responders to Modafinil Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C1538/3048/AD/US
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention-Deficit/Hyper Activity Disorder; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
The purpose of this study is to evaluate the continued efficacy of modafinil treatment, compared to placebo treatment, in children and adolescents with attention-deficit/hyperactivity disorder (ADHD) who are responders to modafinil treatment.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the continued efficacy of modafinil treatment, compared to placebo treatment, in children and adolescents with attention-deficit/hyperactivity disorder (ADHD) who are responders to modafinil treatment, as assessed by the change from baseline (in this current study) in the total score from the ADHD Rating Scale, Fourth Edition (ADHD-RS-IV) (Home Version) at endpoint (week 6 or last double-blind post-baseline visit).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be currently enrolled in a Cephalon-sponsored clinical study and have completed at least 12 months of continuous modafinil treatment. Patients will be included in the study if they continue to meet all applicable criteria in their previous study and all of the following criteria are met:

  * Written informed consent/assent is obtained.
  * The patient is currently enrolled in study C1538d/312/AD/US or C1538/3044/AD/US and received modafinil treatment, continuously, for at least 12 months.
  * The patient meets the protocol criteria for response at each of the last 2 visits of their previous study. Patients from study C1538d/312/AD/US must have at least a 25% reduction in Attention-Deficit/Hyperactivity Disorder Rating Scale - IV [ADHD-RS-IV] (Home Version) total score compared with the original baseline (this must be the baseline for a previous double-blind, placebo-controlled study of modafinil in ADHD). Patients from study C1538/3044/AD/US must have at least a 25% reduction in total score of the ADHD Index subscale of the Conners' Parent Rating Scale: Revised, Short Form (CPRS:R-S), compared with the baseline value from study C1538/3044/AD/US.
  * The patient is in good health (except for diagnosis of ADHD) as determined by medical and psychiatric history, physical examination, electrocardiograms (ECGs), serum chemistry, hematology, urinalysis, and vital signs.
  * Girls who are post-menarche or sexually active must have a negative urine pregnancy test at the baseline visit, must be using a medically acceptable method of birth control, and must agree to continue use of this method for the duration of the study (and for 30 days after participation in the study). Acceptable methods of birth control include the following: barrier method with spermicide; steroidal contraceptive (eg, oral, transdermal, implanted, or injected) in conjunction with a barrier method; intrauterine device (IUD); and abstinence.
  * The patient has a parent or legal guardian who is willing to participate in the study.

Exclusion Criteria:

* Patients are excluded from participating in this study if 1 or more of the following criteria are met:

  * The patient has a history or current diagnosis of pervasive developmental disorder, schizophrenia, or other psychotic disorders, or positive clinical assessment of current suicide risk or ideation.
  * The patient has any current psychiatric co-morbidity that requires pharmacotherapy, including but not limited to depression or other mood disorder, anxiety disorder, or pervasive mental disorder.
  * The patient currently uses any other prescription medication, other than modafinil, for ADHD (eg, amphetamine, dextroamphetamine, methylphenidate, pemoline, atomoxetine).
  * Previous exposure to modafinil caused any clinically significant (drug-related) adverse reaction that led to withdrawal from the study, or which the investigator considers likely to put the patient at risk.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120
Dates: Start 2006-06; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - UCI Child Development Center, Irvine, California
  - University of California at San Francisco, San Francisco, California
  - Encompass Clinical Research, Spring Valley, California
  - Alpine Clinical Research, Boulder, Colorado
  - Sarkis Family Psychiatry, Gainesville, Florida
  - Amedica Research Institute, Inc., Hialeah, Florida
  - Miami Research Associates, Miami, Florida
  - Child Neurology Associates, Atlanta, Georgia
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Michael J. Rieser, MD, PSC, Lexington, Kentucky
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Clinical Neurophysiology Services, Troy, Michigan
  - University of Nebraska, Omaha, Nebraska
  - CNS Research Institute, Clementon, New Jersey
  - Piedmont Neuropsychiatry, Charlotte, North Carolina
  - Triangle Neuropsychiatry, Durham, North Carolina
  - Pahl Pharmaceutical Research, Inc., Oklahoma City, Oklahoma
  - OCCI, Inc., Salem, Oregon
  - The Clinical Study Center, Burlington, Vermont
  - Monarch Research Associates, Norfolk, Virginia
  - Eastside Therapeutic Resource, Kirkland, Washington
  - Pacific Institute Mental Health, Seattle, Washington